CLINICAL TRIAL: NCT01457443
Title: Biomarker for Pompe Disease AN INTERNATIONAL, MULTICENTER, EPIDEMIOLOGI-CAL PROTOCOL
Brief Title: Biomarker for Pompe Disease (BioPompe)
Acronym: BioPompe
Status: Withdrawn | Type: Observational
Why Stopped: Transition into BioMetabol
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: BP 06-2018
Record Dates: First submitted 2011-10-21; First posted 2011-10-24 (Estimated); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Cardiac Diseases; Muscular Weakness; Hepato-splenomegaly; Lung Disease; Obstructive Sleep Apnoea; Macroglossia; Cerebral Aneurysm
Keywords: Pompe Disease; Biomarker
MeSH Terms: conditions — Heart Diseases; Muscle Weakness; Lung Diseases; Sleep Apnea, Obstructive; Macroglossia; Intracranial Aneurysm; Glycogen Storage Disease Type II

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For the development of the new biomarkers using the technique of mass-spectometry, maximal 10 ml blood will be taken from the patient via using a dry blood spot filter card. To proof the correct Pompe diagnosis in those patients where up to the enrollment in the study no genetic testing has been done, sequencing of Pompe will be done as rou-tine diagnostic.
  The analyses will be done at the:
  Centogene AG Am Strande 7 18055 Rostock Germany
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation: Patients with Pompe disease

SUMMARY:
Development of a new MS-based biomarker for the early and sensitive diagnosis of Pompe disease from blood (plasma)

DETAILED DESCRIPTION:
Pompe disease is a rare (estimated at 1 in every 40,000 births), inherited and often fatal disorder that disables the heart and muscles. It is caused by mutations in a gene that encodes an enzyme called alpha-glucosidase (GAA). Normally, the body uses GAA to break down glycogen, the long-term storage form of sugar, into glucose, which the body can utilize to gain energy. But in Pompe disease, mutations in the GAA gene reduce or completely eliminate the activity of this essential enzyme. Excessive amounts of glycogen accumulate everywhere in the body, but the cells of the heart and skeletal muscles are the most seriously affected. Re-searchers have identified up to 70 different mutations in the GAA gene that cause the symptoms of Pompe disease, which can vary widely in terms of age of onset and severity. The severity of the disease and the age of onset are related to the degree of enzyme deficiency.

Early onset (or infantile) Pompe disease is the result of complete or near complete deficiency of GAA. Symptoms begin in the first months of life, with feeding problems, poor weight gain, muscle weakness, floppiness, and head lag. Respiratory difficulties are often complicated by lung infections. The heart is grossly enlarged. More than half of all infants with Pompe disease also have enlarged tongues. Most babies with Pompe disease die from cardiac or respiratory complications before their first birthday.

Late onset (or juvenile/adult) Pompe disease is the result of a partial deficiency of GAA. The onset can be as early as the first decade of childhood or as late as the sixth decade of adulthood. The primary symptom is muscle weakness progressing to respiratory weakness and death from respiratory failure after a course lasting several years. The heart may be involved but it will not be grossly enlarged. A diagnosis of Pompe disease can be confirmed by screening for the common genetic mutations or measuring the level of GAA enzyme activity in a blood sample - a test that has 100 percent accuracy. Once Pompe disease is diagnosed, testing of all family members and consultation with a professional geneticist is recommended. Carriers are most reliably identified via genetic mutation analysis.

New methods, like mass-spectrometry give a good chance to characterize in the blood (plasma) of affected patents specific metabolic alterations that allow to diagnose in the future the disease earlier, with a higher sensitivity and specificity.

Therefore it is the goal of the study to develop new biochemical markers from the plasma of the affected patients helping to benefit the patient by an early diagnose and thereby with an earlier treatment.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent will be obtained from the patient or the parents before any study related procedures.
* Patients older than 12 months
* The patient has a diagnosis of Pompe disease

Exclusion Criteria:

* No Informed consent from the patient or the parents before any study related procedures
* Patients younger than 12 months
* The patient has no diagnosis of Pompe disease

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Pompe disease
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Development of a new MS-based biomarker for the early and sensitive diagnosis of Pompe disease from plasma | 24 month
  New methods, like mass-spectrometry give a good chance to characterize specific metabolic alterations in the blood of affected patients that allow diagnosing in the future the disease earlier, with a higher sensitivity and specificity

SECONDARY OUTCOMES:
Testing for clinical robustness, specificity and long-term stability of the biomarker | 36 months
  the goal of the study to identify and validate a new biochemical marker from the blood of the affected patients helping to benefit other patients by an early diagnose and thereby with an earlier treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bauer, Prof., Study Chair — Centogene GmbH
Locations (4):
- Centogene AG, Rostock, Germany
- India (2):
  - Amrita Institute of Medical Sciences & Research Centre, Kochi, Kerala
  - Navi Mumbai Institute of Research In Mental And Neurological Handicap (NIRMAN), Mumbai
- Lady Ridgeway Hospital for Children, Colombo, Sri Lanka

IPD SHARING:
Plan to Share IPD: Undecided